CLINICAL TRIAL: NCT04820153
Title: Monitoring Physical Activity in Hispanic Women With Chronic Neurological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Giselle Petzinger, MD, Clinical Scholar, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-18-00993
Record Dates: First submitted 2019-01-27; First posted 2021-03-29 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Neurological Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study Participants (Other): Study participants will participate in both the Physical Activity Monitoring Device intervention and the Lifestyle Redesign Coaching intervention simultaneously. Both interventions are complementary to one another.
  Interventions: Device: Physical Activity Monitoring Device; Behavioral: Lifestyle Redesign Coaching

INTERVENTIONS:
Device: Physical Activity Monitoring Device — Participants will be provided a Fitbit Alta HR and wall charger. Each participant will be assigned a unique ID# at baseline and used to set-up the data acquisition. The Fitbit app will be set up on their smartphone to allow self-monitoring of activity. The Fitbit device includes both an accelerometer and heart rate monitor, capable of continuous measuring and storing data up to 5 days. Fitbit data will be passively downloaded through smartphone connection to Fitabase, a research friendly application and data management program. The Fitbit will be worn on the wrist every day during the course of the 16-week study, with instructions on self- monitoring, usage and maintenance. Participants will be monitored for Fitbit compliance by weekly phone calls; and monitoring of passively downloaded Fitbit data through Fitabase. Follow-up phone call at 3-months post-study will assess continued use of the Fitbit activity monitor.
Behavioral: Lifestyle Redesign Coaching — Participants will receive individualized goal setting and a guide to increase exercise at baseline and at week four visit. The Occupational therapist (OT) will administer a well published approach for promoting PA called Lifestyle Redesign which addresses physical, psychosocial and environmental barriers to health and incorporate self-care strategies and goal setting. Coaching will be administered by a bilingual OT and in Spanish. Based on studies examining PA and brain health, the OT will guide the participant through a goal setting process for moderate to vigorous intensity of physical activity including a specific guide plan to achieve these goals of 10,000 steps per day and/or 150 minutes/week of moderate to vigorous activity. Participants will also receive weekly calls from the study coordinator (overseen by OT) to review PA and goal setting for each week over the course of the 16-week study.

SUMMARY:
The primary goal of this proposal is to demonstrate the feasibility of using a Fitbit charge to monitor and promote physical activity in a diverse population of Hispanic women with chronic neurological disorders. Hispanic women will also receive behavioral coaching using a Lifestyle Redesign approach to enhance physical activity in their daily lives. The secondary goal of this proposal is to investigate whether changes in physical activity are associated with (i) quality of life including perception of health and well- being and (ii) frequency of hospital and county clinic visits.

DETAILED DESCRIPTION:
This pilot study will provide feasibility on use of wearable technology for tracking and self-monitoring physical activity (PA) as well as preliminary data to support our overall approach for promoting PA and improving disease status in a Hispanic women population. A larger application will be submitted to the NIH, DoD, or other federal agency focused on investigating the impact of PA on chronic neurological diseases in a diverse and inclusive Hispanic population in LA County.

2.1.1 Specific Aim 1 establishes feasibility of this approach by measuring adherence and change in PA using a Fitbit alta HR activity monitor in Hispanic women with chronic neurological diseases. Adherence will be determined through: (i) the average hours/day of use; and (ii) the length of time (percent of total study days) of usage throughout the 16-week study. Adherence defined as (i) 5 or more days/week of use and (ii) 10 or more hours of use during the day.

2.1.2 Specific Aim 2 tests the hypothesis that an increase in physical activity will be correlated with a decrease in LA County (LAC) Facilities health care use (hospital and clinic visits). Physical activity will be assessed by change in either: (i) the average number of steps/week; and (ii) average time spent in sedentary, light, or moderate to vigorous intensity based on MET (metabolic expenditure) of physical activity/week. Methods: Changes in PA outcome metrics over the 16-week period will be correlated with the total number of hospital/outpatient clinic visits. Total hospital use will be determined through the LAC/DHS (Department of Human Services) electronic medical records and will include outpatient provider visits, emergency room and urgent care visits, total hospitalizations, and days spent in hospital.

2.1.3 Specific Aim 3a tests the hypothesis that increase in physical activity is associated with an increase in the quality of life (QOL). Physical activity will be measured through: (i) the average number of steps/week; and (ii) average intensity of physical activity/week. QOL will be determined through measures of self-rated health and well-being. These Spanish validated surveys will include illness perception questionnaire and health and well-being questionnaire

ELIGIBILITY:
Inclusion Criteria includes

* (1) Women of Hispanic origin;
* (2) established patient of the neurology clinic defined as clinic visits at the LAC/USC Neurology Clinic that have spanned greater than one year;
* (3) age > 30
* (4) willing and able to utilize a Fitbit activity Monitor;
* (5) own a smart phone device;
* (6) ambulatory without assistance;
* (7) willing and able to provide informed consent;
* (8) within commuting distance to the wellness center and LAC/USC hospital;
* (9) reads or comprehends Spanish;
* (10) weekly internet access.

Exclusion Criteria includes

* (1) Clinically significant neurological or psychiatric illness including mental retardation, dementia or severe depression/anxiety;
* (2) any physical condition that precludes engagement in exercise, including significant heart disease.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Baseline Demographic Data | At Baseline Visit
  Baseline demographic data will be obtained which will include age, recent healthcare visit frequency, medical history, medication, years of education, and tobacco use.
Physical Activity Adherence Assessment- Step Count + | 16 weeks
  Data gathered from Fitbit based device will be stored, visualized and aggregated through a commercially available service (Fitabase Inc, Https:/www.Fitabase.com). Step Count will be obtained during the course of the study.
Physical Activity Adherence Assessment- Time spent in moderate to vigorous activity | 16 weeks
  Data gathered from Fitbit based device will be stored, visualized and aggregated through a commercially available service (Fitabase Inc, Https:/www.Fitabase.com).Time spent in moderate to vigorous activity will be obtained during the course of the study.
Physical Activity Adherence Assessment- length of wear. | 16 weeks
  Data gathered from Fitbit based device will be stored, visualized and aggregated through a commercially available service (Fitabase Inc, Https:/www.Fitabase.com). Length of wear will be obtained during the course of the study.
Determination of LA County Facilities Health Care Use- number of inpatient LA County Hospital visits | 16 weeks
  The investigators will utilize electronic medical record (EMR) system of LA County Department of Health Services (DHS) to determine the number of inpatient hospital visits The total number of visits to the LAC/USC medical center will be determined during the 16-week period prior to study initiation and during the period of the study intervention using electronic medical records. HIPPA guidelines will be followed.
Determination of LA County Facilities Health Care Use- number of LA County Hospital Outpatient visits | 16 weeks
  The investigators will utilize electronic medical record (EMR) system of LA County Department of Health Services (DHS) to determine the number of outpatient hospital visits. The total number of visits to the LAC/USC medical center will be determined during the 16-week period prior to study initiation and during the period of the study intervention using electronic medical records. HIPPA guidelines will be followed.

SECONDARY OUTCOMES:
Quality of Life (QOL) Assessment | At Baseline Visit and Week 16
  This measure assessed participants' views of their health, how well they feel, and how well they are able to complete their usual activities. The scale is comprised of 16 items with a 1-7 rating scale of points. A higher sum of points indicates feelings of better quality of life and a better outcome.
Spanish Acculturation | At Baseline
  The purpose of this questionnaire is to assess the level to which participants acculturate or adopt the attitudes, values, customs, beliefs, and behaviors of another culture. The scale is comprised of 12 items measured on a scale of 1 to 5, which are averaged. Low acculturation is measured by an average score >2.99.
Brief Illness Perception Questionnaire (BIPQ) | At Baseline and Week 16
  The purpose of this questionnaire is to assess participants' perceptions of their health and well-being.
  Each item of the Brief IPQ assesses one dimension of illness perceptions:
  The consequences score is simply the response to item 1. The timeline score is the response to item 2 The personal control scores is the response to item 3 The treatment control score is the response to item 4 The identity score is the response to item 5 The coherence score is the response to item 7 The emotional representation is the response to item 8. Illness concern is measured by item 6. This reflects a combination of emotional and cognitive representations.
  Item 9 is the causal item. Reponses can be grouped into categories such as stress, lifestyle, hereditary, etc. determined by the particular illness studied. Categorical analysis can then be performed, either on just the top listed cause or all three listed causes.
Spanish Physical Activity Questionnaire | At Baseline and Week 16
  This self-administered questionnaire determines total physical activity (MET-h week-1 ) and total number of hours sitting down across a week to evaluate the levels of participants' physical activity and sedentary lifestyle. The number of METs (metabolic equivalents) corresponding to each activity are calculated using the Compendium of Physical Activities as the ratio of energy expended during a physical activity to the metabolic rate. Afterwards, the number of METs in each activity is multiplied by the weekly participation in that activity. The estimated number of MET-h week -1 is weighted according to the number of months dedicated to each activity. Recreational physical activity is quantified by summing the MET-h week -1 dedicated to all activities performed during leisure time. Total physical activity (MET-h week -1) is calculated by adding leisure-time physical activity to work physical activity.
FitBit Wear Technology Questionnaire | At Week 16
  The purpose of this questionnaire is to ascertain participants' opinions on the usability of the Fitbit phone application, Fitbit activity monitor, and combination of the Fitbit and Fitbit Application. Participants score questions pertaining to usability on a scale of 1 (strongly disagree) to 5 (strongly agree). These scores are averaged and expressed as a percentage of 100, with higher scores indicating greater usability.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Petzinger, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in the study may contact PI to request information regarding study protocol and de-identified study data.
Supporting Information: Study Protocol
Time Frame: upon completion of study.
Access Criteria: Researchers interested in the study may contact PI to request information regarding study protocol and de-identified study data.

REFERENCES:
- [Derived] Garbin A, Diaz J, Bui V, Morrison J, Fisher BE, Palacios C, Estrada-Darley I, Haase D, Wing D, Amezcua L, Jakowec MW, Kaplan C, Petzinger G. Promoting Physical Activity in a Spanish-Speaking Latina Population of Low Socioeconomic Status With Chronic Neurological Disorders: Proof-of-Concept Study. JMIR Form Res. 2022 Apr 20;6(4):e34312. doi: 10.2196/34312. PMID 35442197

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT04820153/Prot_SAP_000.pdf